CLINICAL TRIAL: NCT03865979
Title: Automated Detection, Characterization, Triage, and Recruitment of ICH Subjects Using Artificial Intelligence in the ENRICH Trial
Brief Title: AI ENRICH - AI Detection of ICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viz.ai, Inc. (Industry)
Collaborators: Nico Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VIZ-ICH-01
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intracerebral Hemorrhage
Keywords: Artificial Intelligence; ICH
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Intervention Arm (Active Comparator): Subject CT images assessed by Viz RECRUIT software in "real time" analysis All subjects in which the Viz RECRUIT software is utilized will be identified per cohort described below per PI confirmation of ENRICH Trial status/Study ID.
  Cohort A: Subjects with imaging data Cohort B: Subjects with imaging data and ultimately enrolled as part of the ENRICH Trial
  Interventions: Device: Viz RECRUIT
- Control Arm (No Intervention): Subjects enrolled as part of the ENRICH Trial prior to Viz RECRUIT software activation

INTERVENTIONS:
Device: Viz RECRUIT — Viz RECRUIT includes the following modules: Viz ICH, Viz VOLUME, Viz VIEW and Viz HUB
  Arms: Intervention Arm

SUMMARY:
To evaluate the performance of the Viz RECRUIT software in subjects identified as symptomatic of a stroke event as determined by standard of care imaging assessments and interpretation.

DETAILED DESCRIPTION:
This study will be a multicenter prospective feasibility trial to evaluate the performance of the Viz RECRUIT software. This study will enroll subjects evaluated at each center for stroke via CT imaging. The Viz RECRUIT software will review the CT and notify a specialist if an ICH is detected. It will also evaluate the ICH parameters per study specific guidelines related to the ENRICH Trial and notify a specialist if their ICH meets the study inclusion or exclusion criteria related to cerebral blood flow volume. If an enrolled subject is ultimately included in the ENRICH trial, they will be identified in a prospective cohort of subjects exposed to Viz (intervention arm) will be evaluated per the secondary endpoints to a cohort of subjects retrospectively from the ENRICH Trial (control arm) which were evaluated and enrolled prior to Viz use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stroke symptoms who undergo CT brain imaging.

Exclusion Criteria:

* Subjects with poor or incomplete CT brain imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Performance | Enrollment
  Rate of concordance of Viz RECRUIT software identification of ICH via Head CT images and standard of care radiologist identification of ICH.

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Jankowitz, MD, Principal Investigator — The Cooper Health System
Locations (6):
- United States (6):
  - UAMS Medical Center, Little Rock, Arkansas
  - Northshore University Health System, Evanston, Illinois
  - Cooper University Hospital, Camden, New Jersey
  - SUNY Buffalo, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Geisinger Medical Center, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No